CLINICAL TRIAL: NCT03714724
Title: The Effects of Various PEEP (Positive End-expiratory Pressure) Levels on Intraabdominal Pressure and Hemodynamics in Critically Ill Patients
Brief Title: PEEP Levels on Intraabdominal Pressure and Hemodynamics in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Assistant professor, Yuzuncu Yil University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PEEP and IAP
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Intraabdominal Hypertension; Critically Ill; Hemodynamic Instability
Keywords: Critically ill patients; intraabdominal pressure; hemodynamics; positive end-expiratory pressure
MeSH Terms: conditions — Intra-Abdominal Hypertension; Critical Illness

STUDY DESIGN:
Intervention Model Description: Intraabdominal pressure of the patients were measured on the 0. 6. 12. 18. and 24. hours and recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 4 (Active Comparator): Patients who received 0-4 cmH2O PEEP in mechanical ventilation were referred to as Group 4.
  Intraabdominal, central venous, arterial blood pressures, pulse rates, peripheric oxygen saturation, body temperature, instant fluid balances and amounts of urine (in ml/kg/hour unit) of the patients were measured on the 0. 6. 12. 18. and 24. hours and recorded.
  Interventions: Diagnostic Test: Intraabdominal Pressure Measurement
- Group 8 (Active Comparator): Patients who received 5-8 cmH2O PEEP in mechanical ventilation were referred to as Group 8. Intraabdominal, central venous, arterial blood pressures, pulse rates, peripheric oxygen saturation, body temperature, instant fluid balances and amounts of urine (in ml/kg/hour unit) of the patients were measured on the 0. 6. 12. 18. and 24. hours and recorded.
  Interventions: Diagnostic Test: Intraabdominal Pressure Measurement
- Group 12 (Active Comparator): Patients who received 9-12 cmH2O PEEP in mechanical ventilation were referred to as Group 12. Intraabdominal, central venous, arterial blood pressures, pulse rates, peripheric oxygen saturation, body temperature, instant fluid balances and amounts of urine (in ml/kg/hour unit) of the patients were measured on the 0. 6. 12. 18. and 24. hours and recorded.
  Interventions: Diagnostic Test: Intraabdominal Pressure Measurement

INTERVENTIONS:
Diagnostic Test: Intraabdominal Pressure Measurement — In this method, a sterile set system (AbViser- Wolfe Tory Medical, Saik Lake City, Utah, USA) was used in normal conditions. Measurements will be made in 20 ml saline was given, Pressure transducer was used as a reset point pubic symphysis and intra-abdominal pressure was measured.

SUMMARY:
In this study, it was aimed to compare the effects of three different PEEP levels (0-4, 5-8, 9-12 cmH2O) on intraabdominal pressure and hemodynamic parameters of patients in intensive care unit.

DETAILED DESCRIPTION:
Patients between 18-80 years old whom were mechanically ventilated without any spontaneous respiratory efforts on supine position were included into the study. Bladder pressure measurement as a practical and frequently preferred method was used in order to measure intra-abdominal pressure. 100 ml isotonic fluid was given during the measurement. Level of symphysis pubis was chosen for zeroing the pressure transducer to measure the intra-abdominal pressure.

Three patient groups, each containing 22 cases, totally 66 patients were planned in this study. All patients were mechanically ventilated with various PEEP levels. The patients with 0-4 cmH2O PEEP levels were named Group 4; the patients with 5-8 cmH2O PEEP levels were named Group 8; the patients with 9-12 cmH2O PEEP levels were named Group 12. The levels of patients' PEEP levels were arranged by the responsible intensive care physician regarding to the patients' clinic.

Intraabdominal, central venous, arterial blood pressures, pulse rates, peripheric oxygen saturation, body temperature, instant fluid balances and amounts of urine (in ml/kg/hour unit) of the patients were measured on the 0. 6. 12. 18. and 24. hours and recorded.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-80,
* connected to mechanical ventilator in intensive care,
* had not undergone surgery of the abdomen,
* patients followed at the same PEEP levels for at least 24 hours

Exclusion Criteria:

* The consent for the study,
* initial intrabdominal pressure level is over 12 cmH2O,
* undergoing abdominal surgery or bladder surgery,
* neurogenic bladder,
* morbid obesity,
* Chronic Obstructive Pulmonary Disease Patients were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
measure intraabdominal pressure | 1 month
  Intraabdominal Pressure Measurement In this method, a sterile set system (AbViser- Wolfe Tory Medical, Saik Lake City, Utah, USA) was used in normal conditions. Measurements will be made in 20 ml saline was given, Pressure transducer was used as a reset point pubic symphysis and intra-abdominal pressure was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yüzkat, Study Chair — Yuzuncu Yil University
Locations (1):
- Van yuzuncu Yıl University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marini M, Caretta G, Vagnarelli F, Luca F, Biscottini E, Lavorgna A, Procaccini V, Riva L, Vianello G, Aspromonte N, Mortara A, De Maria R, Capasso P, Valente S, Gulizia MM. [Hemodynamic effects of positive end-expiratory pressure]. G Ital Cardiol (Rome). 2017 Jun;18(6):505-512. doi: 10.1714/2700.27611. Italian. PMID 28631764
- [Result] Verzilli D, Constantin JM, Sebbane M, Chanques G, Jung B, Perrigault PF, Malbrain M, Jaber S. Positive end-expiratory pressure affects the value of intra-abdominal pressure in acute lung injury/acute respiratory distress syndrome patients: a pilot study. Crit Care. 2010;14(4):R137. doi: 10.1186/cc9193. Epub 2010 Jul 21. PMID 20663183